CLINICAL TRIAL: NCT04822012
Title: Anti COVID-19 Antibodies in Spermatic Fluid and Follicular Fluid
Brief Title: Anti COVID-19 Antibodies in Follicular Fluid and Spermatic Fluid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Anat Hershko Klement, Unit director, Meir Medical Center
Other Study IDs: 0053-21-HMO
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: SARS-CoV-2
Keywords: infertility; SARS-CoV-2,COVID-19
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Follicular fluid post egg retreival and spermatic fluid post fertilization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female: Female patients going through an egg retrival procedure and were identified as post COVID-19 vaccine/ post COVIS-19 infection or not post vaccine/post disease and screened negative for COVID-19 in the week prior to the procedure.
  Interventions: Diagnostic Test: Anti COVID19 IgG Antibodies
- Male: male patients going through an in vitro fertilization cycle and were identified as post COVID-19 vaccine/ post COVIS-19 infection or not post vaccine/post disease and screened negative for COVID-19 in the week prior to the procedure.
  Interventions: Diagnostic Test: Anti COVID19 IgG Antibodies

INTERVENTIONS:
Diagnostic Test: Anti COVID19 IgG Antibodies — Detection of antibodies to SARS Cov 19 post infection or vaccination , measurements of female hormones in folicular fluid as compared to serum and Perlecan as a follicular quality marker
  Other Names: Estrogen and Progesterone levels in serum and follicle; Follicular Perlecan level

SUMMARY:
Patients going through an in vitro fertilization cycle will be asked to participate . Patients will be asked for their COVID-19 exposure : post confirmed disease/post vaccine/not exposed to disease or vaccine . Patients will provide the fluids which are not required , once fertilization process is completed. Patients will also provide 5ml blood sample by the day of procedure. Anti COVID-19 immunoglobulin G type antibodies will be measured in all samples . Data regarding age, date of infection/vaccine will be collected . Progesterone and Estrogen will be measured in female patients' samples and Perlecan level will be measured in follicular fluid.

DETAILED DESCRIPTION:
Patients going through an in vitro fertilization cycle will be asked to participate . Patients will be asked for their COVID-19 exposure : post confirmed disease/post vaccine/not exposed to disease or vaccine . Patients will provide the fluids which are not required in the day of egg retrieval : the follicular fluid remaining after isolation of the egg and spermatic fluid only, if not utilized for fertilization. The fluids will be collected once fertilization process is completed. Patients will also provide 5ml blood sample by the day of procedure. Anti COVID-19 immunoglobulin G type antibodies will be measured in all samples . Data regarding age, date of infection/vaccine will be collected as well as indication for treatment, Estradiol level before the egg retrieval, number of eggs collected and the triggering ovulation modality . Progesterone and Estrogen will be measured in female patients' samples (follicular fluid and serum). Perlecan level will be measured in follicular fluid.

ELIGIBILITY:
Inclusion Criteria:

* Planned egg retrieval procedure (including egg preservation)
* Negative PCR for SARS-Cov-19 in the week before egg retrival
* Informed consent

Exclusion Criteria:

* Positive PCR for SARS-Cov-19 in the week before egg retrival
* expected retrival of 1-3 eggs

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Patients going through an artificial reproductive procedure : females performing egg retrieval and males performing in vitro fertilization with their female partner. Each addressed separately for informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Follicular - Serum Anti COVID-19 antibody (Immunoglobulin G) ratio | Through study completion, expected 2 months
  The relationship between antibodies to COVID-19 in serum to follicular fluid in female patients going through an egg retrieval
Spermatic fluid- Serum Anti COVID-19 antibody (Immunoglobulin G) ratio | Through study completion, expected 2 months
  The relationship between antibodies to COVID-19 in serum to spermatic fluid in male patients going through in vitro fertilization treatment

SECONDARY OUTCOMES:
Follicular fluid Estradiol level (pmol/L) | Through study completion, expected 2 months
  Quality assessment of follicular fluid as measured by Estradiol level
Follicular fluid Progesterone level (nmol/L) | Through study completion, expected 2 months
  Quality assessment of follicular fluid as measured by Progesterone level
Follicular fluid Perlecan level (nmol/L) | Through study completion, expected 2 months
  Quality assessment of follicular fluid as measured by Perlecan level

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Batiha O, Al-Deeb T, Al-Zoubi E, Alsharu E. Impact of COVID-19 and other viruses on reproductive health. Andrologia. 2020 Oct;52(9):e13791. doi: 10.1111/and.13791. Epub 2020 Aug 13. PMID 32790205
- [Background] Segars J, Katler Q, McQueen DB, Kotlyar A, Glenn T, Knight Z, Feinberg EC, Taylor HS, Toner JP, Kawwass JF; American Society for Reproductive Medicine Coronavirus/COVID-19 Task Force. Prior and novel coronaviruses, Coronavirus Disease 2019 (COVID-19), and human reproduction: what is known? Fertil Steril. 2020 Jun;113(6):1140-1149. doi: 10.1016/j.fertnstert.2020.04.025. Epub 2020 Apr 16. PMID 32482250
- [Derived] Bentov Y, Beharier O, Moav-Zafrir A, Kabessa M, Godin M, Greenfield CS, Ketzinel-Gilad M, Ash Broder E, Holzer HEG, Wolf D, Oiknine-Djian E, Barghouti I, Goldman-Wohl D, Yagel S, Walfisch A, Hersko Klement A. Ovarian follicular function is not altered by SARS-CoV-2 infection or BNT162b2 mRNA COVID-19 vaccination. Hum Reprod. 2021 Aug 18;36(9):2506-2513. doi: 10.1093/humrep/deab182. PMID 34364311